CLINICAL TRIAL: NCT00438061
Title: Effect of Weight Loss on Lipoprotein Metabolism in Abdominal Obesity
Brief Title: Effect of Abdominal Obesity on Lipoprotein Metabolism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Western Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC-256
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2007-02-26 (Estimated); Status verified 2007-02

CONDITIONS: Obesity; Dyslipidemia; Insulin Resistance
Keywords: Lipoprotein metabolism; Cardiovascular disease; Obesity
MeSH Terms: conditions — Obesity; Dyslipidemias; Insulin Resistance; Cardiovascular Diseases

INTERVENTIONS:
Behavioral: Weight loss by dietary restriction

SUMMARY:
Abdominal obesity is strongly associated with dyslipidemia, which may account for the associated increased risk of atherosclerosis and coronary disease. Weight reduction is suggested to be a preferred and effective first-line strategy to correct lipid abnormalities, particularly in overweight/obese subjects. This improvement may be related to the effect of reduction in abdominal fat mass on apoB and apoA-I metabolism, but this remains to be fully demonstrated.

Hypothesis: Reduction in abdominal fat mass by weight loss decreases apoB concentration and raises HDL-cholesterol chiefly by increasing LDL-apoB fractional catabolic rate (FCR), as well as decreasing HDL apoA-I, respectively.

DETAILED DESCRIPTION:
We examined the mechanism of the effect of weight loss through dieting on LDL and HDL metabolism in abdominally obese men. LDL apoB-100 and HDL apoA-I kinetics were studied using a primed-constant infusion of 1-[13C]-leucine in a controlled, dietary intervention trial of 16 weeks duration in middle-aged, obese men with the metabolic syndrome. Isotopic enrichment in apoB and apoA-I was measured by gas chromatography-mass spectrometry and fractional turnover rates estimated using multi-compartmental modelling.

ELIGIBILITY:
Inclusion Criteria:

* Obesity was defined as a body mass index (BMI) >28kg/m2 and visceral visceral obesity (waist to hip ratio> 1.0 or waist circumference >100 cm)

Exclusion Criteria:

* Diabetes mellitus,
* Proteinuria,
* Hypothyroidism,
* Abnormal liver enzymes,
* Major systemic illness,
* A history of alcohol abuse,
* A family history of hyperlipidemia or premature coronary artery disease or were taking medication known to affect lipid metabolism.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 1995-01; Study Completion 1998-12

PRIMARY OUTCOMES:
Primary: Fractional catabolic and production rates of LDL-apoB and HDL-apoA-I (before and after 16 week treatments)

SECONDARY OUTCOMES:
Secondary: Cholesterol; Triglyceride; LDL-cholesterol; Adipocytokines; Genetic polymorphism

CONTACTS AND LOCATIONS:
Overall Officials: Dick C Chan, PhD, Principal Investigator — The University of Western Australia; Gerald F Watts, MD, Study Chair — The University of Western Australia
Locations (1):
- Royal Perth Hospital, Perth, Western Australia, Australia